CLINICAL TRIAL: NCT06756490
Title: A Prospective, Blinded (Evaluators and Subjects Blinded), Randomized Controlled Phase I Clinical Trial to Evaluate the Safety, Efficacy and Pharmacokinetics of Liposome-encapsulated Deoxycholic Acid for Injection (HY-2003) Administered by Subcutaneous Fat Layer Injection in the Subjects With Excessive Submental Fat Accumulation
Brief Title: A Phase I Study of HY-2003 in the Subjects With Excessive Submental Fat Accumulation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Huiyu Pharmaceutical Co., Ltd (Industry)
Collaborators: Peking Union Medical College Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HY-2003-101
Record Dates: First submitted 2024-12-17; First posted 2025-01-03 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Moderate or Severe Submental Fullness
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A - Subjects will be randomly assigned to three subgroups (Experimental)
  Interventions: Drug: HY-2003 (10 mg/ml), BELKYRA and placebo
- Group B - Subjects will be randomly assigned to two subgroups (Experimental)
  Interventions: Drug: HY-2003 (5 mg/ml) and placebo
- Group C - Subjects will be randomly assigned to two subgroups (Experimental)
  Interventions: Drug: HY-2003 (5 mg/ml) and placebo

INTERVENTIONS:
Drug: HY-2003 (10 mg/ml), BELKYRA and placebo — Participants received HY-2003 (10 mg/ml), or BELKYRA, or placebo administered up to 10 mL per treatment session at intervals of approximately 4 weeks for up to a maximum of 6 treatments.
  Arms: Group A - Subjects will be randomly assigned to three subgroups
Drug: HY-2003 (5 mg/ml) and placebo — Participants received HY-2003 (5 mg/ml) or placebo administered up to 10 mL per treatment session at intervals of approximately 2 weeks for up to a maximum of 6 treatments.
  Arms: Group B - Subjects will be randomly assigned to two subgroups
Drug: HY-2003 (5 mg/ml) and placebo — Participants received HY-2003 (10 mg/ml) or placebo administered up to 10 mL per treatment session at intervals of approximately 4 weeks for up to a maximum of 6 treatments. It is possible to explore the maximum number of administrations exceeding six treatment sessions.
  Arms: Group C - Subjects will be randomly assigned to two subgroups

SUMMARY:
The main purpose of this study is to evaluate the safety of HY-2003 in subjects with moderate to severe submental fat accumulation at different doses and dosing frequencies in comparison with the positive control and placebo. The secondary objectives include: Evaluating the pharmacokinetic characteristics of HY-2003 after a single administration in humans and obtaining preliminary pharmacokinetic parameters; Evaluating the efficacy of HY-2003 under different doses and dosing frequencies, compared with the positive control and placebo, in the treatment of subjects with moderate to severe submental fat accumulation.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the requirements of the trial, and signed the informed consent form voluntarily;
2. The subjects should have good compliance, are able to fully understand this clinical trial, have reasonable expectations for the injection effects, and can abide by the research procedures until the end of the clinical trial.
3. Aged 18 to 65 years (including boundary values), male or female.
4. At screening and baseline, the investigator rated moderate to severe submental outline protrusion due to submental fat accumulation according to the clinician-reported Submental Fat Rating Scale (CR-SMFRS), i.e., those with a score of 2 to 3 points.
5. Sufficient submental fat to allow for safe subcutaneous fat layer injections (at least 25 injections can be completed), as judged by the investigator.
6. Stable body weight for at least 6 months prior to Screening.
7. Vital sign examinations, physical examinations, clinical laboratory examinations (blood routine, urine routine, blood biochemistry, infectious disease screening, coagulation function, pregnancy test (for females), drug screening, etc.), and 12-lead electrocardiogram examinations, with the results showing no abnormalities or having abnormalities but judged by the researcher as being of no clinical significance.
8. Subjects had no pregnancy plans and voluntarily take effective contraceptive measures during the screening period and within 6 months after the last dose, and have no sperm or egg donation plans.

Exclusion Criteria:

1. Subjects who have previously undergone surgical operations, liposuction treatments in the submental area that may affect the implementation and/or evaluation of the study, or have been injected with lipolytic drugs similar to the study drugs (for example, phosphatidylcholine, etc.).
2. Subjects who have had previous allergic reactions to deoxycholic acid or other components of the investigational drug.
3. History of hypersensitivity to topical or local anesthetics (e.g., lidocaine, benzocaine, procaine, etc.).
4. Subjects with a history of prior surgery in the chin or neck region; or significant submental scarring, infection, cancerous or precancerous lesions, and/or unhealed wounds, mandibular retrusion (a mandibular retrusion malocclusion caused by mandibular hypoplasia or congenital absence of lower anterior teeth and lateral pterygoid insufficiency) that could affect the evaluation results as assessed by the investigator.
5. Subjects with chin and neck skin diseases, or with a keloid-forming tendency (with a previous tendency of scar hyperplasia or keloid), which may affect the efficacy evaluation or subject safety as judged by the investigator.
6. Subjects who have received previous lipolytic therapy with poor efficacy or serious adverse reactions.
7. Platissimus muscle protrusion at rest, as judged by the investigator, impacts assessment of submental fat status.
8. Including but not limited to Madelung's disease (benign symmetric lipomatosis) which leads to an increase in local fat in the neck area and needs to be excluded as judged by the investigator.
9. Body Mass Index (BMI) less than 17 or greater than 40 kg/m2 (excluding borderline) at screening.
10. Current or past dysphagia.
11. Subjects with very severe laxity of the submental skin as judged by the investigator.
12. Enlargement of the submental area was found to be due to other causes rather than local excessive submental fat accumulation.
13. Subjects who have used drugs that can prolong the clotting time (for example, aspirin, non-steroidal anti-inflammatory drugs, clopidogrel, warfarin, etc.) within 2 weeks before screening, or who need to take any drugs with anticoagulant functions (including but not limited to warfarin, heparin) during the trial.
14. Subjects who have used topical drugs (such as glucocorticoids, tretinoin ointment) on the submental skin within 1 month before screening, or who are expected to need to use these drugs on the submental area during the research process (until 12 weeks after the completion of the last injection).
15. Subjects who have donated blood (including blood components) or suffered from massive blood loss (≥200 mL) within 3 months before screening.
16. Subjects who smoked more than 5 cigarettes per day within 3 months before screening, or who were unable to stop using any tobacco products during the PK blood sampling period.
17. Subjects who consumed more than 14 units of alcohol per week within 3 months before screening (1 unit of alcohol is approximately equivalent to 360 mL of beer, 45 mL of spirits with an alcohol content of 40%, or 150 mL of wine), or who were unable to abstain from alcohol during the PK blood sampling period.
18. Subjects who consumed any food or beverage containing caffeine or that can produce caffeine after metabolism (such as coffee, tea, chocolate) within 48 hours before drug administration; or those who did not agree to refrain from consuming such food or beverage during the PK blood sampling period.
19. Subjects who participated in any other drug clinical trials and received drug treatment within 3 months before screening.
20. Subjects with a history of drug abuse within 6 months before screening or who used drugs within 3 months before screening.
21. Subjects who received ultrasonic scalpel, radiofrequency, laser surgery, chemical peeling or skin fillers (such as hyaluronic acid) treatment for the neck or submental area within 12 months before screening, or who received botulinum toxin injection treatment for the neck or submental area within 6 months before screening; or who received non-invasive skin tightening treatment within 6 months before screening.
22. According to the researcher's judgment, the dissolution of submental fat would cause submental skin laxity or have other anatomical features (for example, protrusion of the subplatysmal fat, skin laxity in the neck or chin area, protrusion of the platysma band), resulting in an unacceptable cosmetic effect.
23. At the time of enrollment screening, the results of coagulation function tests, including prothrombin time (PT) and activated partial thromboplastin time (APTT), showed bleeding abnormalities of clinical significance.
24. Subjects who cannot tolerate venipuncture, have a history of fainting due to needles or blood, or have significant abnormal clinical manifestations.
25. Subjects with diseases that require exclusion due to significant abnormal clinical manifestations, including but not limited to diseases of the nervous system, cardiovascular system, blood and lymphatic system, immune system, kidneys, liver, gastrointestinal tract, respiratory system, metabolism, skeletal system and other systems.
26. Subjects suffering from any diseases that may interfere with the safety assessment of the trial or affect the normal conduct of the clinical trial by the subjects or the signing of the informed consent form.
27. Subjects whose participation in the trial may increase their risks or who may have other severe, acute or chronic diseases that may interfere with the interpretation of the trial results and are judged by the researcher as not suitable for participating in the clinical trial.
28. Subjects who plan to undergo any surgeries or take any drugs that may lead to significant changes in body weight (≥10%) during the study period (for example, systemic corticosteroids, weight-loss drugs, bariatric surgeries).
29. Subjects with infectious diseases before screening, such as syphilis, AIDS, hepatitis B, etc.
30. Female subjects with potential fertility who are pregnant, breastfeeding, planning to become pregnant or not taking reliable contraceptive measures, and who are unwilling to adopt reliable contraceptive methods (for example: transdermal patches, intrauterine devices/systems (IUD/IUS), oral/implanted or injected contraceptives, abstinence and vasectomy of their spouses) during the participation in the trial.
31. Subjects with other comorbidities that may interfere with the research assessment only as judged by the researcher, or subjects who are considered by the researcher as facing greater risks due to participation in the study.
32. Subjects judged by the researcher as not suitable for participating in this trial for other reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-26 (Actual); Primary Completion 2026-02-05 (Estimated); Study Completion 2026-02-05 (Estimated)

PRIMARY OUTCOMES:
The occurrence of all adverse events; The occurrence of adverse events at the injection site; Laboratory tests, vital signs, physical examinations, 12-lead electrocardiograms. | During the intervention
Pain scores evaluated by the Visual Analogue Scale (VAS，0~10mm，the longer the length means a worse outcome） | During the intervention
The scores of submental skin laxity evaluated by the Submental Skin Laxity Grade (SMSLG, 0~4 points, the higher score means a worse outcome） | Four weeks and twelve weeks after the last treatment.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: No